CLINICAL TRIAL: NCT06432270
Title: A Prospective Cohort Study of the Effect of Diabetes Mellitus on Cardiac Autonomic Function in Surgical Patients Undergoing General Anesthesia
Brief Title: Effect of Diabetes Mellitus on Cardiac Autonomic Function in Surgical Patients Undergoing General Anesthesia
Status: Not yet recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-KY-209-02
Record Dates: First submitted 2024-05-07; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Autonomic Neuropathy Type 2; Perioperative Complication; Temperature Change, Body
Keywords: diabetes; general anesthesia; Cardiac autonomic dysfunction; perioperative temperature
MeSH Terms: conditions — Body Temperature Changes; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic group: Patients with a diagnosis of diabetes mellitus who are about to undergo general anesthesia who are expected to undergo laparoscopic surgery
- Non-diabetic group: Nondiabetic patients anticipating laparoscopic surgery who are about to undergo general anesthesia

SUMMARY:
Because autonomic neuropathy affects the constriction of thermoregulatory blood vessels, it is more difficult for diabetic patients to maintain their own body temperature in cold environments than normal people, and therefore it is more difficult for diabetic patients to maintain a relatively constant body temperature regardless of the temperature of the environment than normal people. So are diabetic patients under general anesthesia more susceptible to intraoperative hypothermia? How does heart rate variability change in diabetic patients under general anesthesia? If diabetic patients are more susceptible to intraoperative hypothermia under general anesthesia, is this related to their cardiac autonomic dysfunction?

DETAILED DESCRIPTION:
According to the latest version of data released by the International Diabetes Federation (IDF) in 2021, it can be seen that the number of people with diabetes globally or in China is high and the percentage is increasing.In 2021, there are 537 million people with diabetes globally, and there are about 141 million in China, which is an increase of about 21.55% compared with 2019 . Perioperative hypothermia is a clinical phenomenon in which a patient's core body temperature is below 36°C for non-medical purposes during the perioperative period, with an incidence of about 7-90%, which can lead to a variety of adverse outcomes.In hot environments, sweating and vasodilation are severely compromised in diabetic patients due to autonomic neuropathy, which prevents the body from transferring heat from the inside of the body to the skin through vasodilation, increased blood flow, and sweating. Similarly, because autonomic neuropathy affects the constriction of thermoregulatory blood vessels, it is more difficult for diabetic patients to maintain their own body temperature in cold environments than normal people, and therefore it is more difficult for diabetic patients to maintain a relatively constant body temperature regardless of the temperature of the environment than normal people. On the other hand, general anesthesia and external environmental factors in the operating room increase the incidence of intraoperative hypothermia, and theoretically, diabetic patients are more prone to dramatic fluctuations in their own body temperature during surgery, making it difficult for them to adapt to changes in the external environment. Due to the complex pathophysiological mechanism of diabetes, which affects multiple systems throughout the body, there are currently more than 100 complications of diabetes, of which autonomic neuropathy has the most serious impact on diabetic patients. Cardiac autonomic neuropathy is one of the most common and serious complications of diabetic autonomic neuropathy, with a prevalence of 63% . And heart rate variability is one of the most common tests for diabetic cardiac autonomic dysfunction. So are diabetic patients under general anesthesia more susceptible to intraoperative hypothermia? How does heart rate variability change in diabetic patients under general anesthesia? If diabetic patients are more susceptible to intraoperative hypothermia under general anesthesia, is this related to their cardiac autonomic dysfunction? However, there are still no studies and little attention has been paid to it.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age ≤ 80 years old, gender is not limited;
* BMI index of 18-35 kg/m2 (including 18 kg/m2 and 35 kg/m2 );
* Diagnosed with diabetes mellitus;
* ASA Ⅰ - Ⅱ;
* Elective laparoscopic abdominal surgery under general anesthesia;
* Operating time >2 hours and <6 hours;
* Voluntary participation and signing of an informed consent form;
* Ability to be followed up in a timely manner.

Exclusion Criteria:

* Abnormally elevated preoperative inflammatory indicators;
* Core body temperature ≥37.5 degrees Celsius;
* Patients with previous clear central nervous system disease, history of psychiatric disorders, or epilepsy;
* Patients with verbal communication or hearing or visual impairment, who were unable to communicate well and had poor compliance;
* Intraoperative use of vasodilator (uradil, sodium nitroprusside, nitroglycerin);
* Any high-risk subjects with complete atrioventricular block or complete atrioventricular conduction tissue without implanted pacemakers, multiple premature ventricular beats, single premature ventricular beats (heart rate <45 beats/min), heart failure in NYHA (New York Heart Association) class III or higher;
* Subjects with any other clinically significant 12-lead electrocardiogram (ECG) or echocardiogram abnormality at the time of screening, ejection fraction (EF) <40%, or any other significant abnormality in the opinion of the investigator;
* Subjects deemed by the investigator to be unfit for this clinical trial for any other reason (anesthesia assessment unfit for surgery or preanesthetic hypertension).

Withdrawal Criteria:

* Serious adverse events, abnormal laboratory tests, or other conditions that indicate no further benefit or increased risk to the subject's safety from continued participation in the study;
* Incomplete recording of critical data (temperature or heart rate variability);
* Unstable condition requiring further admission to the intensive care unit;
* Intraoperative use of dexmedetomidine; 5. Perioperative nerve block.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is expected to collect patients who are hospitalized in Zhujiang Hospital of Southern Medical University and are proposed to undergo surgery
Sampling Method: Non-Probability Sample
Enrollment: 388 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in perioperative core body temperature in diabetic patients | 12 hours before surgery,during operation,12 hours after surgery
  The study was conducted by using a perioperative core body temperature monitoring system to continuously monitor and record core body temperature data for 12 hours preoperatively - intraoperatively - 12 hours postoperatively, and then calculating the mean core body temperature per minute at 12 hours preoperatively, intraoperatively, and 12 hours postoperatively, respectively, to compare whether diabetic patients had lower mean core body temperature per minute intraoperatively than non-diabetic patients, and whether diabetic patients had a decrease in intraoperative body temperature compared to 12 hours preoperatively and 12 hours postoperatively. Mean intraoperative core body temperature per minute (°C/min) = Mean intraoperative core body temperature/operating time.

SECONDARY OUTCOMES:
time to onset of temperature drop | Baseline and 12 hours before surgery,0-30 minutes after induction ,30-60 minutes after induction,60-90 minutes after induction,90-120 minutes after induction,120-150 minutes after induction,150-180 minutes after induction,12 hours after surgery
  observing the time period during which diabetic and non-diabetic patients began to drop below the mean temperature at 12 hours preoperatively and comparing how early or late the temperature began to drop in both groups
time to temperature drop to nadir | Baseline and 12 hours before surgery,0-30 minutes after induction ,30-60 minutes after induction,60-90 minutes after induction,90-120 minutes after induction,120-150 minutes after induction,150-180 minutes after induction,12 hours after surgery
  Observing the period of time during which diabetic and non-diabetic patients experienced a drop in temperature to nadir, and comparing how fast or slow the temperature dropped to the lowest point
The magnitude of body temperature decline | Baseline and 12 hours before surgery,0-30 minutes after induction ,30-60 minutes after induction,60-90 minutes after induction,90-120 minutes after induction,120-150 minutes after induction,150-180 minutes after induction,12 hours after surgery
  Comparing whether the average core body temperature of diabetic patients was lower than that of non-diabetic patients at each time period after induction.
Changes in heart rate variability (HRV) | 12 hours before surgery,12 hours after surgery
  using 24-hour Holter ECG to collect HRV data from 12 hours before surgery to induction (first administration of medication), and from the time the patients left the recovery room to 12 hours after surgery, and observing the changes in HRV data of the patients of the two groups in the two time periods

OTHER OUTCOMES:
Age | the preoperative visit period
  Age of the participants(years)
Height | the preoperative visit period
  Height of the participants(meters)
BMI | the preoperative visit period
  BMI of the participants(kg/m2)

CONTACTS AND LOCATIONS:
Overall Officials: Zhujiang Hospital of Southern Medical University, Study Chair — Southern Medical University, China

IPD SHARING:
Plan to Share IPD: Undecided